CLINICAL TRIAL: NCT02471872
Title: Behavioral Research of Environment and Air Pollution Through Education (BREATHE Study)
Brief Title: Behavioral Research of Environment and Air Pollution Through Education
Acronym: BREATHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mehrdad Arjomandi, Professor of Medicine in the Division of Pulmonary, Critical Care, Allergy, Immunology, and Sleep Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BREATHE
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Attitude to Health; Pollution Related Respiratory Disorder; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air Pollution Education (Experimental): Students are presented with a one-hour interactive information session about air pollution and the environment.
  Interventions: Behavioral: Air Pollution Education
- Non-Air Pollution Education (Placebo Comparator): Students are presented with a one-hour interactive information session about vaccines.
  Interventions: Other: Non-Air Pollution Education

INTERVENTIONS:
Behavioral: Air Pollution Education — Students are presented with a one-hour interactive session on air pollution.
  Arms: Air Pollution Education
Other: Non-Air Pollution Education — Students are presented with a one-hour interactive session on vaccines.
  Arms: Non-Air Pollution Education

SUMMARY:
The BREATHE (Behavioral Research of Environment and Air Pollution Through Education) study is a pilot randomized control trial comparing the efficacy of a classroom-based intervention to no intervention in helping middle-school students understand and make behavioral decisions about air pollution. This study is designed to evaluate the effectiveness of the classroom-based intervention on knowledge of air pollution, understanding of air pollution sources, and behavioral choices made to reduce both contributions to air pollution and personal exposure to air pollution.

It has been well established that pollution is a racial and economic issue. Low-income areas with populations of predominantly people of color tend to be those with the highest rates of pollution and the largest particulate exposure. Creation of and exposure to this pollution is a key issue for the health of inhabitants of these areas, and of those in the broader surrounding areas. By developing, and assessing the effectiveness of, the investigators hope that the BREATHE study will give the investigators insights into how to better combat this higher exposure and reduce the health risks for those in high pollution areas.

The study will take place in 4 visits over a period of 12 months. The hypothesis is that the classroom-based intervention will be effective in leading to behaviors that will reduce exposure to air pollution.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, write, and understand English at a middle school level
* Willing to participate in follow up visits

Exclusion Criteria:

* Learning disabilities such as autism
* Moving out of the area in the next 6 months
* Inability to complete the questionnaires

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Behavior Change Assessed by Questionnaires | Assessed immediately after intervention, and at 3 months, 6 months, and 12 months
  Change in Future Behavior as it Relates to Personal Choices and Support for Policies and Regulations

SECONDARY OUTCOMES:
Improvement in Understanding Assessed by Questionnaires | Assessed immediately after intervention, and at 3 months, 6 months, and 12 months
  Improvement in Understanding of Air Pollution and Its Public Health Ramification

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided